CLINICAL TRIAL: NCT00489372
Title: Phase I Study of Single Oral Dose of Se-Methyl-Seleno-L-Cysteine (MSC) in Adult Men
Brief Title: Se-Methyl-Seleno-L- Cysteine (MSC) in Treating Healthy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2013-00505; NCI-2013-00505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 87406; NCI04-4-02; NWU04-4-02 (Other: Northwestern University); NWU04-4-02 (Other: DCP); P30CA060553 (NIH); N01CN35157 (NIH)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-09

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — selenomethylselenocysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (placebo) (Placebo Comparator): Participants receive oral placebo on day 1.
  Interventions: Other: placebo; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (Se-methyl-seleno-L-cysteine) (Experimental): Participants receive oral Se-methyl-seleno-l-cysteine (MSC) on day 1. Cohorts of 5 participants receive escalating doses of MSC until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 5 or 2 of 10 patients experience dose-limiting toxicity.
  Interventions: Drug: Se-methyl-seleno-L-cysteine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Se-methyl-seleno-L-cysteine — Given orally
  Other Names: methylselenocysteine; MSC
  Arms: Arm II (Se-methyl-seleno-L-cysteine)
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm I (placebo)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of Se-methyl-seleno-L-cysteine in healthy adult men. Studying samples of blood, urine, and toenail clippings in the laboratory from healthy men receiving Se-methyl-seleno-L-cysteine may help doctors learn more about how Se-methyl-seleno-L-cysteine works in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity of MSC, given to healthy adult males as a single oral dose.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of single oral doses of MSC in healthy adult male volunteers.

II. To evaluate the baseline selenium content of toenail clippings in healthy adult males.

OUTLINE: This is a multicenter, randomized, placebo controlled, double blind, dose escalation study. Participants are randomized to 1 of 2 arms.

Arm I: Participants receive oral placebo on day 1.

Arm II: Participants receive oral Se-methyl-seleno-l-cysteine (MSC) on day 1. Cohorts of 5 participants receive escalating doses of MSC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 or 2 of 10 patients experience dose-limiting toxicity.

Participants undergo blood, urine, and toenail clipping collection for pharmacokinetic and correlative studies. Samples are analyzed for plasma protein levels of selenium for proteomic and gene expression, molecular fingerprinting by mass spectrometry, and RNA by gene array analysis.

After completion of study treatment, participants are followed at 7-14 days and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Total body weight between 50 and 115 kg
* Hgb > 12 gm/dl
* Platelets > 100,000/μL
* ANC > 1000/μL
* Creatinine < 1.5 mg/dl
* SGPT and SGOT < 3 X the institutional upper limit of normal (ULN)
* Total bilirubin < 1.5 X the institutional ULN (subjects with a higher level of bilirubin due to a familial metabolism will be considered on an individual basis)
* Life expectancy greater than 2 years
* Male subjects must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and until study completion (i.e., at least two weeks after dose of study drug)
* Ability to understand and the willingness to sign a written informed consent document
* Agree to refrain from use of selenium supplements while on study

Exclusion Criteria:

* Not willing to remain at RPCI, and in follow up, as required
* Presence of medical conditions, which in the opinion of the investigators, would compromise either the subject, or the integrity of the data
* Individuals with a history of active liver or kidney disease within the past 6 months
* Treatment with an investigational drug within 30 days prior to the dose of study drug
* Use of prescription or nonprescription drugs, vitamins, or herbal supplements known to change gastric acidity (e.g., H2-antagonists, proton pump inhibitors, antacids) within 3 days of study drug administration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MSC (e.g. reaction to other selenium supplements)
* Subjects who have donated 1 unit of blood within 30 days prior to the first dose of MSC
* Subjects with a known history of heavy metal exposure, such as lead, mercury, of arsenic
* ECOG performance status > 1
* AUA total symptom score > 10 (or any individual symptom score of greater than or equal to 4 will exclude the participant)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Clinical toxicity in healthy adult male volunteers, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v3.0 | Up to 30 days
  Summarized using descriptive statistics.

SECONDARY OUTCOMES:
Characterization of the pharmacokinetics of MSC | Up to 24 hours post-dose
  Descriptive statistics calculated for each cohort, using established pharmacokinetic analysis methods.
Selenium levels in toenail samples | Up to 24 hours post-dose
  Summarized graphically.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Bergan, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York